CLINICAL TRIAL: NCT06788496
Title: RCT Pilot Study: Art-based Beauty Appreciation Intervention
Brief Title: Art-based Beauty Appreciation Intervention
Acronym: ABBA-vention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Amsterdam (Other); University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL87597.091.24
Record Dates: First submitted 2024-12-22; First posted 2025-01-23 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-12

CONDITIONS: Young Adults; Sensory Processing Sensitivity
Keywords: Beauty Appreciation; Well-being; Mental Health; Young Adults; Active Control Condition; Art Based Intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Masking Description: The researchers were also blind to the randomization block size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Control Condition (Active Comparator)
  Interventions: Behavioral: Observation Program (Learning to Observe Life)
- Intervention Condition (Other)
  Interventions: Behavioral: Art-based Beauty Appreciation Intervention Program (Learning to See Beauty)

INTERVENTIONS:
Behavioral: Art-based Beauty Appreciation Intervention Program (Learning to See Beauty) — The goals of the intervention program are to help individuals develop an aesthetic mindset, practice observation and appreciation skills, learn how to apply these skills to their day-to-day lives, practice emotion regulation with beauty, and incorporate more beauty into their lives. The program is designed to create a slow skill transfer from appreciation in art contexts to natural beauty and to everyday life. In the 14-day program, participants visit an art museum with guided audio, watch instructional videos about observing and appreciating beauty, and complete daily written or photo beauty journals that document the beauty they see. In addition, participants will watch video art showing how to find beauty in mundane objects, practice this in a beauty walk, and complete a planning session to include more beauty in their lives.
  Arms: Intervention Condition
Behavioral: Observation Program (Learning to Observe Life) — The active, matched control group will focus on developing pragmatic observation skills. Participants will be instructed to pay attention to and identify objects and elements in their surroundings without emphasizing their aesthetic value. For example, they should pay attention and count objects of the same colour they encounter, social behaviour, the people they pass on the street, or the types of buildings. The 14-day program includes a tourist trip with guided audio instruction, watching instructional videos about increasing observation skills and completing daily written or photo journals to document their observations. Further, participants will take an observation walk and plan to include more observation in their lives.
  Arms: Active Control Condition

SUMMARY:
This study is a randomized controlled trial with an active control condition evaluating the impact of an art-based beauty appreciation (ABBA) intervention on trait appreciation of beauty as a primary outcome and well-being and psychological distress as secondary outcomes. The central hypothesis is that the primary and secondary outcomes will increase more in the intervention than in the control condition.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with an active control condition evaluating the impact of an art-based beauty appreciation (ABBA) intervention on trait appreciation of beauty as a primary outcome and well-being and psychological distress as secondary outcomes. These two programs have been designed and validated in a qualitative pilot study as matched in credibility, intensity, and enjoyment. There are three measurement points for primary and secondary outcomes, including (1) enrollment, (2) a post-test after the intervention/control program, and (3) a 4-week follow-up measure. N = 114 participants will be randomized after baseline into either the intervention or control group (N = 57/group). In addition, to investigate perceived mechanisms, barriers, and facilitators, participants will be selected using purposive sampling and invited to a semi-structured interview until data saturation is reached (expected N = 15).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between 18-28 years of age,
2. indicate that they have a smartphone to support our data collection and program components,
3. have the ability and interest to make a trip to a museum or new location (i.e., new part of the city),

(3) be willing to complete short activities every day for two weeks, (4) and be fluent in English, (6) be based in Amsterdam, (7) are willing to share postal address to receive materials.

Exclusion Criteria:

1. Participants must not currently be in clinical treatment for a mental health disorder, assessed via self-report, or
2. indicate that they are currently experiencing severe psychological symptoms (i.e., depression, suicidal ideation, severe anxiety) via self-report.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Engagement with Beauty | From baseline to the follow-up period (up to 2 months)
  The Engagement with Beauty Scale Revised (EBS-R) is an 18-item self-report scale designed to assess cognitive and emotional engagement with natural beauty, artistic beauty, moral beauty, and beautiful ideas. Participants respond on a 7-point Likert scale, ranging from 1 (very unlike me) to 7 (very much like me). Example items include reflections on physiological responses to natural beauty, the spiritual experience elicited by art, and the desire for personal growth through moral beauty appreciation. Subscales measure engagement with moral beauty (scores 6-42) and the other three domains (scores 4-28), contributing to a total score ranging from 18 to 126.

SECONDARY OUTCOMES:
Well-being | From baseline to the follow-up period (up to 2 months)
  We will measure well-being using the Mental Health Continuum Short Form (MHC-SF). This has 14 items over three subscales: emotional well-being, social well-being (eudemonic well-being), and psychological well-being. The items are scored on a 6-point Likert scale (0-5), then sum-scored.
Psychological Distress | From baseline to the follow-up period (up to 2 months)
  The DASS-21 will be used to measure psychological distress. It has 21 items divided over three subscales of 7 items each. These capture emotional states of depression, anxiety, and stress. The items are assessed using a four-point Likert scale (0-3), summed together, and multiplied by two. This results in three subscales and a total score.

OTHER OUTCOMES:
Emotion Regulation via Beauty | From baseline to the follow-up period (up to 2 months)
  The Emotion Regulation Strategies for Artistic Creative Activities Scale (ERS-ACA; Fancourt et al., 2019) will be used with slight modification to the question stem. While the initial purpose of this scale was geared towards creative pursuits, it has been rooted in the principles of emotion regulation theory and designed to be applied to various activities. We anticipate that it will be a valuable instrument in evaluating how appreciating beauty can regulate emotions. This change in the question stem concerns the use of the prompt, "When I am appreciating beauty…". Items can be added up to avoidance strategies (i.e., I can block out unwanted thoughts or feelings), approach strategies (i.e., it makes me reflect on my emotions), and self-development strategies (i.e., it reaffirms my identity).
Attention Regulation | From baseline to the follow-up period (up to 2 months)
  Attention regulation will be assessed using the 20-item Attention Control Scale (ACS) (Derryberry & Reed, 2002). The questionnaire consists of 2 subscales: (1) Attention Focusing and (2) Attention Shifting. The items are assessed on a four-point Likert scale (1-4) and will be sum-scored.
Mindfulness Skills | From baseline to the follow-up period (up to 2 months)
  Mindfulness will be assessed using the Five Facet Mindfulness Questionnaire Short Form (FFMQ-15), with 15 items (Baer, Carmody, & Hunsinger, 2012), with five facets: (1) observing, (2) describing, (3) acting with awareness, (4) non-judging, and (5) non-reactivity (Baer et al., 2006). The items are assessed on a five-point Likert scale (1-5) from rarely to always. Scores will be summed for each facet and the total score.
Burnout | From baseline to the follow-up period (up to 2 months)
  Burnout will be measured using the Burnout Assessment Tool-12 (BAT-12), consisting of 12 items (Redelinghuys & Morgan, 2023; Schaufeli et al., 2020). This questionnaire measures burnout with four subscales: (1) Exhaustion, (2) Mental Distance, (3) Emotional Impairment, and (4) Cognitive Impairment (Schaufeli et al., 2020). The items are assessed on a five-point Likert scale (1-5). A total score can be obtained by calculating all items' average scores. Additionally, subscale scores are obtained by calculating the average of the items per subscale.
Qualitative Interview | After timepoint 3 (8-9 weeks after enrollment)
  Semi-structured interview focusing on the impacts of intervention, mechanisms, barriers and facilitators.

CONTACTS AND LOCATIONS:
Overall Officials: MacKenzie D Trupp, PhD Candidate, Study Director — RadboudUMC, Donders Institute for Brain, Cognition and Behaviour and University of Vienna; Corina Greven, Prof. Dr., Principal Investigator — RadboudUMC, Donders Institute for Brain, Cognition and Behaviour
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All identifying information will remain in storage within the RadboudUMC storage systems at the Donders Institute and will not be shared. Data will not be published; however, it will be stored in the Radboud Repository, where further researchers can request access to pseudonymized data after signing a data-access agreement.
Supporting Information: SAP
Time Frame: The study pre-registration will be embargoed on Open Science Framework (OSF) until the publication of the results in an academic journal.
Access Criteria: After the release from the embargo, anyone can access the pre-registration on OSF.